CLINICAL TRIAL: NCT01411449
Title: Drug Use Investigation of EOB-Primovist Inj. Syringe
Brief Title: Primovist Post-marketing Surveillance in Japan
Acronym: PRIMOVIST
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15040
Record Dates: First submitted 2011-08-05; First posted 2011-08-08 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Diagnostic Imaging
Keywords: Primovist; MRI agent
MeSH Terms: interventions — gadolinium ethoxybenzyl DTPA

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Gadoxetic Acid Disodium (Primovist, BAY86-4873)

INTERVENTIONS:
Drug: Gadoxetic Acid Disodium (Primovist, BAY86-4873) — Patients who will need to undergo contrast enhanced MRI with Primovist

SUMMARY:
This study is a regulatory post marketing surveillance in Japan, and it is a local prospective and observational study of patients who have received Primovist for contrast enhancement in MRI of liver. The objective of this study is to assess safety, especially in relation to renal dysfunction, and efficacy of using Primovist in clinical practice. A total 2,000 patients for diagnosis on detection and identify hepatic tumor will be recruited and followed 7 days after the injection.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received Primovist for liver MRI

Exclusion Criteria:

* Patients who are contraindicated based on the product label

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population of this study is patients who received Primovist for liver MRI. The study is expected to collect data of 2,000 patients in about 150 hospitals in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 2030 (Actual)
Dates: Start 2008-03-11 (Actual); Primary Completion 2010-12-14 (Actual); Study Completion 2015-02-18 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions and serious adverse events in subjects who received Primovist | After Primovist injection, up to 7 days
Incidence of adverse drug reactions in patients with renal impairment | After Primovist injection, up to 7 days

SECONDARY OUTCOMES:
Incidence of adverse drug reactions in subpopulation in a variety of baseline data [such as demographic data, concomitant disease and dose of Primovist] | After Primovist injection, up to 7 days
MRI image evaluation assessment by the five rank scales of 1 to 5: 1) much improved; 2) improved; 3) slightly improved; 4) not improved; and 5) impaired | After Primovist injection, up to 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Japan